CLINICAL TRIAL: NCT01073410
Title: Chitinases and TGFB in Human Asthma
Brief Title: Chitinases and Transforming Growth Factor Beta (TGFB) in Human Asthma
Acronym: AADCRC
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 10-02173; U19AI077439 (NIH)
Record Dates: First submitted 2010-02-19; First posted 2010-02-23 (Estimated); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — sputum, blood, saliva, DNA, RNA, Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy, non-asthmatic controls: People who are non-asthmatic and non-smokers.
- Asthmatics: People who have been diagnosed with asthma.

SUMMARY:
The purpose of this study is to find out the roles of two specific gene families (the chitinase gene family and the TGFB family). We hypothesize that chitinases and TGFb pathway genes will be differentially expressed in the airways of non-asthmatic subjects and subjects with asthma. We further hypothesize that genetic variants in CHIT1, AMCase, and TGFb pathway genes that show associations with asthma and related phenotypes will change the expression and/or function of the protein of these genes in the airway in several ways, including the transcript numbers for full length genes and splice variants and, for the chitinase genes, the levels of chitinase activity in airway secretions.

DETAILED DESCRIPTION:
This is a cross-sectional study in patients with asthma and healthy controls in which we will analyze how the expression or function of CHIT1, AMCase, and TGFb pathway genes in the asthmatic airway is affected by genetic variation in these genes. We propose detailed phenotyping of the asthmatic subjects and the healthy controls, including collection of induced sputum, exhaled air and detailed physiologic measures including measures of airflow, lung volumes, and methacholine responsiveness as well as collection of airway cells and tissues by bronchoscopy. We will determine the relative expression of CHIT1 and AMCase in specific lung compartments (large airways, small airways, epithelial cells, macrophages) and the effects of genetic variants in CHIT1 and AMCase on expression of splice variants and levels of chitinase activity in the airway. These human samples will also allow us to determine if any of the multiple TGFb pathway genes analyzed show differential expression in the lung in asthma.

ELIGIBILITY:
Inclusion Criteria:

* History of asthma
* No use of oral or inhaled corticosteroids for the treatment of asthma in the past 6 weeks
* Hyperreactivity to methacholine (PC20FEV1 Methacholine ≤ 8.0 mg/mL).
* At least one of the following symptoms, beta agonist use, or FEV1 criteria:

  * Asthma symptoms on at least two days per week, or
  * Beta agonist use on at least two days per week, or
  * FEV1 < 85% predicted
* Subjects must be non-smokers (patients who have never smoked or patients who have not smoked for 1 year and have a total pack-year smoking history < 10 packs).

Exclusion Criteria:

* Cigarette smoking: Subjects must be non-smokers. Non smokers are defined as subjects who have never smoked or who have not smoked for 1 year and have a total pack-year smoking history < 10 packs.
* Pregnant women
* Subjects with a history of a medical disease which in the opinion of the investigator may put the subject at extra risk from study-related procedures or because the disease may influence the results of the study.
* Healthy control subjects must have no history of asthma or allergic rhinitis
* Upper respiratory tract infection in the 4 weeks prior to enrollment in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2010-02; Primary Completion 2017-02 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
Expression of CHIT1, AMCase, and TGFb pathway genes in asthma | Current

CONTACTS AND LOCATIONS:
Overall Officials: John G Fahy, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Airway Clinical Research Center, San Francisco, California, United States